CLINICAL TRIAL: NCT05054153
Title: Westlake Precision Nutrition Study: Diet Challenges for Glucose Metabolism
Brief Title: Westlake Precision Nutrition Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20210802ZJS001
Record Dates: First submitted 2021-08-24; First posted 2021-09-23 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2021-08

CONDITIONS: Healthy; Overweight and Obesity
Keywords: Glucose Metabolism; Intermittent fasting; Personalized Nutrition; Brain; Gut Microbiome
MeSH Terms: conditions — Overweight; Obesity; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- refined carbohydrate breakfast (Breakfast A) (Experimental): white bread (50g) + milk powder (25g)
  Interventions: Other: refined carbohydrate breakfast
- whole grain breakfast (Breakfast B) (Experimental): plain oats (35g) + milk powder (25g)
  Interventions: Other: whole grain breakfast
- intermittent fasting (IF) (Experimental)
  Interventions: Other: intermittent fasting

INTERVENTIONS:
Other: refined carbohydrate breakfast — After wearing CGM on Day 1, participants will be provided with breakfast A once daily on Day 2, Day 5 and Day 6. Breakfast A contains white bread (50g) and milk powder (25g). Since lunch and dinner would serve as wash-out meals, participants will be free to choose food but provide a record of their diets.
  Other Names: Breakfast A
  Arms: refined carbohydrate breakfast (Breakfast A)
Other: whole grain breakfast — After wearing CGM on Day 1, participants will be provided with Breakfast B once daily on Day 3, Day 4 and Day 7. Breakfast B contains plain oats (35g) and milk powder (25g). Since lunch and dinner would serve as wash-out meals, participants will be free to choose food but provide a record of their diets.
  Other Names: Breakfast B
  Arms: whole grain breakfast (Breakfast B)
Other: intermittent fasting — The period during Day 8 to Day 13 is intermittent fasting period. Participants will experience the moderate fasting on Day 9 and Day 12, which means their daily energy intake is expected to be controlled within 500-600 kcal limit. In these two days, participants will be provided with all three meals. Percentages of macronutrients of provided meals will follow the Recommended Dietary Health guidelines for Chinese residents. The oral glucose tolerance test (OGTT) will be conducted in the morning on Day 8 and Day 13, to test short-term impact of IF intervention on individuals' glucose tolerance. The breakfasts on Day 10 and Day 11 will be the same as that in fasting days. Other meals will be wash-out meals.
  Other Names: IF
  Arms: intermittent fasting (IF)

SUMMARY:
This is a dietary intervention study, which aims to explore different diet challenges for glucose metabolism, including carbohydrates and intermittent fasting (IF) dietary pattern. Considering the glucose responses to the same food are largely heterogeneous among people, this study integrates the concepts of precision nutrition and N-of-1 design. The study also aims to explore differences in brain structure and function between participants with different Body Mass Index (BMI) from the perspective of gut-brain axis.

DETAILED DESCRIPTION:
This study aims for precision nutrition. Participants will be required to wear continuous glucose monitoring (CGM) for 14 days. The diet intervention will be carried out after wearing CGM on Day 1. Individual N-of-1 trial design will be employed during Day 2 to Day 7 to compare the difference of postprandial glucose response to white bread or plain oats. These two breakfasts will appear in alternating order every successive 2 days, and these successive 2 days will be defined as one set. There will be 3 sets during Day 2 to Day 7. Between lunch and dinner will be the wash out period for the remaining effect of the last breakfast intervention on blood glucose homeostasis. In this period, participants will be allowed to choose foods without restrictions, but dietary records are required. The period during Day 8 to Day 14 is defined as intermittent fasting (IF) period, and participants will experience moderate fasting on Day 9 and Day 13 with total energy intake restrained within 500-600 kcal. In these two fasting days, participants will be provided with daily three meals. Investigators will closely monitor participants' latent adverse response and compliance to ensure the intervention will be completed with adequate safety and high compliancy. Oral glucose tolerance test (OGTT) will be conducted in the morning of Day 8 and Day 14 to test the changes of glucose tolerance before and after one set of IF intervention. Electroencephalogram (EEG) and functional Magnetic Resonance Imaging (fMRI) scanning will be conducted as per standard procedure at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Participants reside in Hangzhou
* Participants have no traveling plans within 3 months

Exclusion Criteria:

* Refusing or unable to give informed consent
* Participants with chronic gastrointestinal diseases and take daily relevant medications
* Participants with metabolic diseases including diabetes, hypertension and cardiovascular diseases (CVD)
* Participants with craniocerebral trauma, cancer, liver disease, kidney disease, or other critical illness, or history of operation or medication
* Participants with bulimia nervosa, post-traumatic stress disorder (PTSD), chronic anxiety and depression or other critical neuronal disorder or history of relevant medication
* Being or to be pregnant or lactating.
* Participants with history of alcohol or drug addiction, or smoke above 15 cigarettes per day
* Concurrently participating other clinical trials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose profiling | 14 days
  Real-time blood glucose fluctuations will be recorded by CGM.
Change of glucose tolerance before and after intermittent fasting | Day 8 and Day 13
  Oral glucose tolerance test will also be conducted.

OTHER OUTCOMES:
Changes of fecal and urine metabolomics profiling | Day 1, Day 8 , Day 11 and Day 14
  Fecal and urine metabolite extracts will be analyzed by performing liquid chromatography/quadrupole time-of-flight mass spectrometry (LC/Q-TOF/MS).
Changes of serum metabolomics profiling | Day 1, and Day 14
  Targeted metabolomics are analyzed based on serum.
Changes of interleukin-1β (IL-1β), IL-6, IL-12 | Day 1, and Day 14
  Serum inflammatory factors (including IL-1β, IL-6, and IL-12) will be tested by enzyme-linked immunosorbent assay (ELISA) in pg/mL.
Changes of tumor necrosis factor-α (TNF-α) | Day 1, and Day 14
  Serum level of TNF-α will be tested by ELISA in ng/mL.
Changes of serum dopamine | Day 1, and Day 14
  Dopamine will be analyzed by serum.
Changes of serum 5-hydroxytryptamine | Day 1, and Day 14
  5- hydroxytryptamine will be analyzed by serum.
Changes of serum gamma-aminobutyric acid | Day 1, and Day 14
  Gamma-aminobutyric acid will be analyzed by serum.
Changes of lipid metabolism | Day 1, and Day 14
  Triglyceride, cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol, apolipoprotein A1 and apolipoprotein B.
Changes of weight | Day 1, Day 8 , Day 11 and Day 14
  Weight will be measured in kilograms.
Height | Day 1
  Height will be measured in centimeters.
Body composition | at enrollment
  Body composition (fat mass, lean mass in kg ) are assessed by bioelectrical impedance analysis.
Changes of both systolic and diastolic blood pressure | Day 1, Day 8 , Day 11 and Day 14
  Both systolic and diastolic blood pressure will be measured in mmHg.
Electroencephalograph(EEG) N2 and P3 amplitudes | at enrollment
  Event-related potentials (N2 and P3 amplitudes) of brain will be assessed by EEG in μV.
Brain images | at enrollment
  Brain structure and function was measured by brain magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhang K, Fu Y, Gou W, Miao Z, Tian Y, Liang Y, Liang X, Shuai M, Xiao C, Wang J, Xu F, Jiang Z, Gao C, Ma S, Ordovas JM, Zheng JS. Quantification of personalized glycemic sensitivity to food and its potential for precision nutrition in a series of n-of-1 trials. Am J Clin Nutr. 2025 Aug;122(2):502-512. doi: 10.1016/j.ajcnut.2025.04.015. Epub 2025 Jun 19. PMID 40754388